CLINICAL TRIAL: NCT04723368
Title: AED-delivery Using Drones in Suspected Out-of-hospital Cardiac Arrest
Brief Title: AED-delivery Using Drones in Suspected OHCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: SOS Alarm Sverige AB (Unknown); Everdrone AB (Unknown); Vastra Gotaland Region (Other Government); Aviation capacity resources AB (ACR) (Unknown); Castellum AB (Unknown)
Responsible Party: Principal Investigator, Andreas Claesson, RN, Associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SS1
Record Dates: First submitted 2021-01-18; First posted 2021-01-25 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Drone; AED; OHCA; EMS; Dispatch centre; UAV
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Automated flying Drone carrying an Automated external defibrillator (AED) (Experimental): Five drone systems are setup to be deployed in suspected OHCA cases as a complement to EMS. This is a single-arm intervention evaluating time benefit of drone delivery of AEDs in suspected OHCA.
  Interventions: Device: Automated flying Drone carrying an Automated external defibrillator (AED)

INTERVENTIONS:
Device: Automated flying Drone carrying an Automated external defibrillator (AED) — Totally n=5 drones are equipped with automated external defibrillators (AEDs). These drones are deployed by the dispatch centre to cases of suspected out-of-hospital cardiac (OHCA) as a complement to standard care (ambulance/EMS) over up to 14 months during daytime Monday to Sunday 08:00-22:00. The bystander onsite receives instructions from the dispatcher to retrieve the AED outside the house when it has been delivered by the drone. The bystander attaches the AED to the patients chest to facilitate early defibrillation.

SUMMARY:
Time to defibrillation is the most important predictor of survival in cardiac arrest. Traditional emergency medical system response is often to slow. The overall aim of this pilot study is to evaluate if drones can deliver Automated external defibrillators (AEDs) to the scene of suspected out-of-hospital cardiac arrest (OHCA) prior to ambulance arrival with clinically relevant time benefits.

DETAILED DESCRIPTION:
This is an observational, non-randomized single group assignment study with the primary purpose of evaluating proportion of AED-delivery prior to ambulance arrival and time benefits.

Totally, five AED-equipped drones will be placed in hangars at five different sites covering a geographic area of about 200 km2 and approximately 125,000 inhabitants for dispatch to suspected cases of OHCA as a complement to standard care i.e., ambulance. By coordinating the operations with local Air Traffic Control (ATC), the risk of airspace conflicts, or in worst case collisions, is mitigated to an acceptable level.

The investigators estimate to enroll some 80 alerts and 60 participants during a study period of up to 14 months. The investigators will closely follow and study the potential of delivering AEDs prior ambulance arrival and timesaving effects as compared to ambulance during a period of up to 14 months in which the investigators will follow and study the potential of delivering AEDs prior ambulance arrival and timesaving effects as compared to ambulance.

The drone operator, Everdrone, has integrated all software and hardware for the concept on the DJI Matrice 600 Pro drone. Examples of added features: an integrated Parachute Rescue System (validated by independent third party using the ASTM F3322 - 18 standard), a high precision sense and avoid system and a winching device to safely lower the AED to ground at delivery. Furthermore, Everdrone AB has fully integrated their system and operational routines with the dispatch central, emergency medical services and aviation organizations. As a result from the previous study (version 1.0) a number of hardware and software improvements have been made to the system (version 2.0):

Five hangars will be setup at optimal locations in each of the five administrative areas. Hangars are large isolated tents 4x4 meters in where the drone is placed, remotely operated and surveiled by camera. Hangars are within fenced areas so that the public has no access. They are equipped with weather stations and an automated gate which automatically will open on alert.

When an emergency 112-call is answered it is indexed by the dispatcher depending on the patients condition. If an OHCA is suspected, the dispatcher indexes the event as a)"ongoing cardio-pulmonary resuscitation (CPR)" or b) "Unconscious with abnormal or absent breathing". If an emergency call is identified within administrative areas AND indexed as "a" or "b" an automated (not manual as with ambulance alerts) alert is sent via radio-alert to the drone operator. This triggers:

* boot-up of the drone
* drone hangar gate opening
* route-planning of the mission
* weather condition confirmation
* remote pilot acceptance of the mission
* remote pilot calling ATC for takeoff approval

The drone system receives an alert from the dispatch center and the drone takes off from the hangar after approval from the drone pilot. For safety reasons all beyond visual line of sight (BVLOS) flights are done within the controlled airspace of Säve airport approval from ATC granted for every single flight. Each flight will be carried out at 60-80 meters of altitude, have a preliminary maximum flight speed of 70 km/h, and a maximum range of 6 km one-way. The drone system is remotely deployed and surveiled from the drone operating center at Everdrone Säve Airport, the drone is dispatched alongside ambulance as a complement to standard care. The drone systems are designed to operate in dry conditions with median winds not exceeding 8 m/s and primarily during daylight conditions.

The AED used is an ultra-light AED (FRED Easyport from Schiller), weighting totally 800 grams with basket and siren. Upon arrival onsite the basket with the AED will be winched down from about 30 m altitude and delivered within 10 meters from the object i.e., the front door or onsite in public areas. Local AED drone support after completed mission includes electrode change battery test, potentially pic-up up the drone after dispatch by the Everdrone personnel.

Dispatch of the drone in suspected OHCA cases will be executed as a complement to standard care i.e., ambulance between 21 April to 1 June 2022, totally up to 14 months of full-scale real-life flights to suspected OHCA victims. Based on historical data of OHCA from the Swedish register for cardiopulmonary resuscitation (SRCR) and first ever dispatch of AED-equipped drones during 2020 the drone systems will be alerted in an estimated 80 cases (about 3.5 flights/ week) of suspected OHCA over the study period. In about 25% of cases, predefined exclusion criteria (rain, median wind > 8 m/s, high rise buildings >20m, pre-flight checklists not OK) will presumably prohibit flights, thus making an estimated 60 cases eligible for inclusion (i.e., drone takes off to deliver AEDs in suspected OHCA.)

For more details about the methods please see the research protocol.

ELIGIBILITY:
Inclusion Criteria:

* All suspected OHCA during 112-calls including drowning
* Within prespecified administrative areas (excluding no delivery- and no-fly zones)
* Hours of operation: 08:00-22:00 (daylight conditions)
* Drone system online

Exclusion Criteria:

Pre-alert:

* Children <8 years
* Trauma
* EMS-witnessed cases

Post alert:

* ATC non-approval of flight
* Rain, winds exceeding 8m/s (median)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion (%) of AED-drone arrival prior to ambulance. | Up to 14 months
  In all alerts of suspected OHCA where a drone took off, comparisons will be done on proportion (%) of AED-drones arriving first on scene vs the proportion (%) of ambulances arriving first on scene.
  Accurate completion of mission is defined as delivery of an AED onsite on the ground in close connection from the OHCA and drone operator reporting arrival status "F" back to the dispatch centre. AEDs shall be accessible to the bystander through T-CPR instructions given by the dispatcher.

SECONDARY OUTCOMES:
Median time difference (min:sec) between AED-drone and ambulance. | Up to 14 months
  In all alerts of suspected OHCA where a drone took off, analysis of time benefit will be done in all cases when the AED-drone arrived first to the scene of a suspected OHCA.
  Median time difference (min:sec) between AED-drone and ambulance will be measured.
  Accurate completion of mission is defined as delivery of an AED onsite on the ground in close connection from the OHCA and drone operator reporting arrival status "F" back to the dispatch centre. Time benefit will be presented overall (% > 3minutes) as well as in continuous data intervals i.e. proportions in: 0-1 min, 1-2 min, 2-3 min, 3-4 min.
c) Proportion (%) of attached drone delivered AEDs prior the arrival of EMS. Percentages. | Up to 14 months
  In all alerts to suspected OHCA where a drone took off, a bystander retrieves the drone delivered AED as instructed in T-CPR protocol by the calltaker and attaches it to the patient before ambulance arrival. Percentages.
d) Proportion (%) of cases defibrillated when a drone delivers an AED before ambulance arrival (real OHCA) | Up to 14 months
  In all alerts to suspected OHCA where a drone took off, a bystander attached the AED to the patient as instructed in T-CPR protocol by the calltaker and administers a shock before ambulance arrival. Percentages.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Resuscitation science, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schierbeck S, Nord A, Svensson L, Ringh M, Nordberg P, Hollenberg J, Lundgren P, Folke F, Jonsson M, Forsberg S, Claesson A. Drone delivery of automated external defibrillators compared with ambulance arrival in real-life suspected out-of-hospital cardiac arrests: a prospective observational study in Sweden. Lancet Digit Health. 2023 Dec;5(12):e862-e871. doi: 10.1016/S2589-7500(23)00161-9. PMID 38000871